CLINICAL TRIAL: NCT03197662
Title: Phase 2 Study: Intranasal Oxytocin vs. Placebo for the Treatment of Hyperphagia in Children and Adolescents With Prader-Willi Syndrome
Brief Title: Intranasal Oxytocin vs. Placebo for the Treatment of Hyperphagia in Prader-Willi Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eric Hollander (Other)
Responsible Party: Sponsor-Investigator, Eric Hollander, Director, Autism and Obsessive Compulsive Spectrum Program and Professor, Department of Psychiatry and Behavioral Sciences, Montefiore Medical Center
Organization: Montefiore Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-8076; FD-R-005106-01 (Other Grant/Funding Number: FDA-OOPD)
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Prader-Willi Syndrome; Hyperphagia
Keywords: Prader-Willi Syndrome; Hyperphagia
MeSH Terms: conditions — Prader-Willi Syndrome; Hyperphagia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Intranasal Oxytocin (IN-OXT) (Experimental): Syntocinon (synthetic oxytocin) will be used in this protocol. Each subject will receive a dose of 16 IU QD ("quaque die" or once a day) and will be instructed to inhale 2 puffs per nostril (4 IU each).
  Interventions: Drug: Intranasal Oxytocin (IN-OXT)
- Placebo Comparator: Matched Placebo (Placebo Comparator): Each subject will receive a dose of 16 IU QD, and will be instructed to inhale 2 puffs per nostril (4 IU each).
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin (IN-OXT) — Each subject will receive a dose of 16 IU QD, and will be instructed to inhale 2 puffs per nostril every day (4 IU each). If needed, treatment will be titrated due to side effects or non-response.
  Other Names: Syntocinon
  Arms: Experimental: Intranasal Oxytocin (IN-OXT)
Drug: Matched Placebo — Each subject will receive a dose of 16 IU QD, and will be instructed to inhale 2 puffs per nostril every day (4 IU each). If needed, treatment will be titrated due to side effects or non-response.
  Arms: Placebo Comparator: Matched Placebo

SUMMARY:
This study is a phase 2 randomized double blind 8-week treatment trial of intranasal OXT vs. placebo in 50 subjects aged 5 to 17 years with PWS in order to assess IN-OXT's affect on measurements of (1) eating behaviors (2) repetitive behaviors (3) weight and body composition (4) quality of life (5) salivary OXT and hormone levels (including ghrelin, pancreatic polypeptide, peptide YY, Glucagon-Like Peptide-1 (GLP-1), insulin, glucagon, testosterone, and estrogen). If superior to placebo, this data will add to the current knowledge that OXT is an effective treatment for hyperphagia as well as other symptoms of PWS.

Funding Source- FDA OOPD

DETAILED DESCRIPTION:
Prader-Willi Syndrome (PWS) is a rare neurodevelopmental disorder caused by lack of expression of paternally derived imprinted material on chromosome 15q11-q13. PWS is characterized by mild to moderate intellectual disabilities, repetitive/compulsive behaviors and rigidity, social cognition deficits and severe hypotonia at birth, followed by the onset of hyperphagia later in life. Obesity is responsible for the majority of the morbidity and mortality associated with PWS, and compulsive eating behaviors are most responsible for diminishing the quality of life for caregivers and family members. Oxytocin has been implicated in the pathophysiology of PWS and there have been small studies of intranasal oxytocin (IN-OXT) in this population. To date, however, studies have not been adequately powered to detect significance in target symptoms of hyperphagia and associated symptoms of individuals with PWS. The primary goal of this study is to examine the safety and efficacy of IN-OXT on hyperphagia, as measured by the Hyperphagia Questionnaire-Clinical Trails, from baseline to week 8. Currently, there are no effective treatments available to manage hyperphagia in patients with PWS.

STUDY DESIGN: This is an 8-week double-blind, randomized study in 50 children with PWS aged 5-17. Participation involves 2 in-person visits to our program and 5 remote visits. Travel expenses will be reimbursed to participating families.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female pediatric outpatients aged 5 to 17 years
2. Must be in PWS nutritional phase 2b or 3 as determined by PI
3. Must be on growth hormone treatment and have been receiving stable doses of growth hormone treatment for at least 3 months prior to screening date. Treatment cannot have been interrupted for more than one week within 3 months of screening.
4. Diagnosis of PWS confirmed by patient medical records.
5. A score of at least moderate severity on the Hyperphagia Questionnaire for Clinical Trials at both screening and baseline visits.
6. Stable dosages of hormone treatments (including testosterone and estrogen supplements) for 4 weeks prior to randomization and for the duration of the study.
7. Stable dosages of metabolic treatments that could affect appetite (including metformin) for 4 weeks prior to randomization and for the duration of the study.
8. Physical exam and laboratory results that are within the normal range for individuals with PWS.
9. Presence of a parent/caregiver/guardian that is able to consent for their participation and complete assessments regarding the child's development and behavior change throughout the study.

Exclusion Criteria:

1. Exposure to any investigational agent in the 30 days prior to randomization.
2. Child not receiving growth hormone treatment
3. Children weighing less than 40 lbs
4. Children with unstable Type 2 Diabetes confirmed by Hemoglobin A1C levels at screening
5. Children with unstable medical co-morbidities at baseline.
6. Children with active upper respiratory infections at screening.
7. A primary psychiatric diagnosis other than Autism Spectrum Disorder (ASD), including bipolar disorder, psychosis, schizophrenia, Post-traumatic stress disorder (PTSD) or major depressive disorder (MDD). These patients will be excluded due to potential confounding results.
8. Pregnant or lactating patients or patients who will not agree to use a double barrier method of contraception. IN-OXT has not been studied in pregnant or lactating women.
9. Females using an estrogen-based contraceptive. As an alternative to an estrogen based contraceptive, subjects will be counseled to use progesterone-based contraceptives; cervical cap; cervical sponges; or spermicidal foam in combination with a condom. Subjects will need to use a double barrier method to be in the study.
10. A medical condition that might interfere with the conduct of the study, confound interpretation of study results or endanger the subject's well-being.
11. A known diagnosis of Rett's Syndrome of Childhood Disintegrative Disorder or marked sensory impairment such as deafness or blindness.
12. Subjects who have changes in allied health therapies, behavioral or educational interventions within four weeks prior to randomization other than those associated with school holidays.
13. Subjects who have had changes in medications or medication doses of risperidone, aripiprazole, other antipsychotic medications, clonidine, guanfacine, stimulants or anti-convulsants within four weeks of randomization.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight (8) study participants who consented were not enrolled as they did not meet inclusion/exclusion criteria (screen failures) or withdrew prior to randomization into the study.
Period: Overall Study
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Started | 15 | 17
Completed (The 2 withdrawals (by family on behalf of their child) took place at baseline after randomization and at ~ Week 2.) | 15 | 15
Not Completed | 0 | 2
Not completed — Withdrawn by family | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Intranasal Oxytocin (IN-OXT): Syntocinon (synthetic oxytocin) will be used in this protocol. Each subject will receive a dose of 16 IU QD and will be instructed to inhale 2 puffs per nostril (4 IU each).
  Intranasal Oxytocin (IN-OXT): Each subject will receive a dose of 16 IU QD, and will be instructed to inhale 2 puffs per nostril every day (4 IU each). If needed, treatment will be titrated due to side effects or non-response.
- Total: Total of all reporting groups
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Customized [Count of Participants; unit: Participants]
  5-6 years old | 2 | 5 | 7
  7-12 years old | 12 | 10 | 22
  13-18 years old | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black/African American | 0 | 0 | 0
  Native Hawaiian/Pacific Islander | 0 | 0 | 0
  White | 12 | 13 | 25
  Multiracial | 2 | 3 | 5
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32
Height [Mean (Standard Deviation); unit: centimeters] — Height (in centimeters) is summarized and reported by study arm using basic descriptive statistics. Population: Data was missing or unable to be collected from 2 participants in the matched Placebo arm including 1 participant who withdrew from the study following randomization.
  centimeters
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 135.6 (16.3) | 130.4 (18.9) | 133.0 (17.6)
Body Weight [Mean (Standard Deviation); unit: kilograms] — Participant body weight, in kilograms, was obtained during baseline visits using a regularly calibrated scale. Body weights are summarized by study arm using basic descriptive statistics. Population: Data was unable to be collected from 1 participant in the matched Placebo arm who withdrew from the study following randomization.
  kilograms
    number analyzed (Participants) | 15 | 16 | 31
    (all) | 40.8 (17.9) | 45.2 (34.9) | 43.1 (26.9)
Body Composition [Median (Full Range); unit: percentage of fat] — Body composition, in particular body fat, will be assessed at baseline via bioelectrical impedance analysis (BIA). Body fat percentage results are summarized and reported by study arm using basic descriptive statistics. Population: Data was missing or unable to be collected from 3 participants the Intranasal Oxytocin arm and 7 participants in the matched Placebo arm including 1 participant who withdrew from the study following randomization.
  percentage of fat
    number analyzed (Participants) | 12 | 10 | 22
    (all) | 20.6 [13.7 to 46.6] | 27.0 [21.5 to 44.3] | 23.5 [13.7 to 46.6]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] — BMI was calculated at baseline using height and weight recordings and reported in kg/m^2. Height recordings in centimeters were converted to meters prior to calculating. BMI results are summarized by study arm using basic descriptive statistics. Population: Data was missing or unable to be collected from 1 participant in the Intranasal Oxytocin arm and 1 participant in the matched Placebo arm who withdrew from the study following randomization.
  kg/m^2
    number analyzed (Participants) | 14 | 16 | 30
    (all) | 20.2 [15.2 to 34.1] | 18.8 [15.9 to 49.0] | 19.5 [15.2 to 49.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Efficacy of Peptide Intranasal Oxytocin (IN-OXT)
Description: Change in efficacy of peptide IN-OXT as measured by changes in hyperphagia from baseline will be assessed using the Hyperphagia Questionnaire for Clinical Trials (HQ-CT). HQ-CT is a caregiver-rated assessment comprised of 9-items that measures the frequency and intensity of hyperphagic behaviors, over the preceding two weeks, in participants with Prader-Willi Syndrome (PWS). The HQ-CT total score is created by summing the 9 item-level responses (ranging from 0 to 4) for a possible range of 0-36 with higher scores indicate more extreme hyperphagia. For purposes of this outcome measure, negative scores represent a decrease in hyperphagia from baseline and positive scores represent an increase in hyperphagia from baseline.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: Data was unable to be collected from 2 participants in the matched Placebo study arm who withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | -6.08 (5.65) | -6.64 (5.05)

2. Secondary Outcome: Change in Repetitive Behavior
Description: Change in Repetitive Behavior from baseline was determined using the Repetitive Behavior Scale Revised (RBS-R) score. The RBS-R is a 44-item form used to measure the full spectrum of repetitive behavior of participants. The child's parent will choose a score that describes how much of a problem the behavior has been over the last month on a 4-point scale ranging from 0 ("Behavior does not occur") to 3 ("Behavior occurs and is severe problem"). The final question asks participants to "lump together" all behaviors described in the RBS-R, and provide a rating (0-100) for how much of a problem these repetitive behaviors are overall: 1 ("Not a problem at all") to 100 ("As bad as you can imagine"). For purposes of this outcome, a change in group mean score from baseline is summarized. A negative score is indicative of a decrease in the frequency and severity of behavioral problems; whereas, a positive score is indicative of an increase in the frequency and severity of behavioral problems.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: Data was unable to be collected from 2 participants in the matched Placebo study arm who withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | -13.2 (14.4) | -8.53 (8.89)

3. Secondary Outcome: Change in Rigid Behavior
Description: Change in Rigid Behavior from baseline was assessed using the Montefiore-Einstein Rigidity Scale-Revised-Prader-Willi Syndrome (MERS-R-PWS). The MERS-R-PWS is designed to assess 3 domains of rigid behavior in children with PWS: 1. Behavioral Rigidity (e.g., insistence on sameness, things must be done his/her way, etc.) 2. Cognitive Rigidity (e.g., special interests, inflexible adherence to rules, etc.) 3. Protest (in response to deviation from rigidity (e.g., verbal objection, tantrum, physical aggression). Four items are rated on a 5-point scale ranging from 0 ("No/None") to 4 ("Extreme/Extremely difficult") for each of the 3 domains. The domains are added yielding a possible Total Domain Score which could range from 0-48. For purposes of this outcome measure, a change in group mean score from baseline is summarized. A negative score is indicative of a decrease in rigid behaviors from baseline; whereas, a positive score is indicative of an increase in rigid behavior from baseline.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: Data was unable to be collected from 2 participants in the matched Placebo study arm who withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | -8.43 (5.15) | -11.2 (7.86)

4. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline was determined by obtaining the participant's body weight, in kilograms, using a regularly calibrated scale. Change in body weights from baseline are summarized by study arm using basic descriptive statistics. A negative result indicates a decrease in body weight from baseline and may be associated with improved health-related outcomes including a decrease in hyperphagia.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: Data was missing or unable to be collected from 3 participants in the matched Placebo study arm (including the 2 participants who withdrew from the study).
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 15 | 14
kilograms | 0.585 (0.709) | -0.0669 (2.14)

5. Secondary Outcome: Body Composition
Description: Body composition, in particular fat mass, was assessed using bioelectrical impedance analysis (BIA). BIA was conducted with equipment and oversight provided by the Einstein-Mount Sinai Diabetes Research Center. The equipment measured resistance in ohms which represents the resistance to a small alternating current passing through the body. These values are converted to body fat percentages using built-in software, after calibrating for variables, for purposes of reporting. Percentages are summarized by study arm using basic descriptive statistics.
Time Frame: 8 weeks
Population: Data was missing or unable to be collected from 4 participants in the IN-OXT study arm and 8 participants in the matched Placebo study arm (including the 2 participants who withdrew from the study).
Measure: Median (Full Range); unit: percentage of fat
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 11 | 9
percentage of fat | 23.5 [15.0 to 53.7] | 24.3 [18.2 to 43.4]

6. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI from baseline will be calculated by dividing the participant's weight in kilograms by their height in meters squared (kg/m^2). Change in mean BMI from baseline will summarized and reported using basic descriptive statistics. A negative BMI score may be indicative of a decrease in hyperphagia from baseline; whereas, a positive BMI score may be indicative of an increase in hyperphagia when compared to baseline.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: Data was missing or unable to be collected from 1 participant in the IN-OXT arm and 3 participants in the matched Placebo study arm (including the 2 participants who withdrew from the study).
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 14 | 14
kg/m2 | 0.229 (1.26) | -0.357 (0.911)

7. Secondary Outcome: Change in Quality of Life (QOL) and Caregiver Burden as Determined by the World Health Organization Quality of Life (WHOQOL-BREF) Questionnaire: Domain 1 (Physical Health)
Description: Change in QOL/Caregiver burden was assessed using the 7-item Physical Health domain subscale of the WHOQOL-BREF questionnaire. The questionnaire was completed by the parent/caregiver and quantified the burden placed on the caregiver/family by the PWS disorder. Each item of the Physical Health domain was scored on a 5-point ordinal scale ranging from 1-5, for an overall possible raw scoring range of 7-35. A mean overall Physical Health score was calculated by summing the scores from the seven items (response values for 2 of the items are inversely-coded) and dividing by the total # of questions (7) for an algebraic mean. A transformed scale score was obtained by subtracting 7 (lowest possible score) from the raw score and dividing by 28 (possible raw score range). For purposes of this outcome measure change from baseline was reported. Increases in Physical Health scores from baseline were associated with higher physical health QOL and reduced caregiver physical burden.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | -0.0714 (2.89) | -0.929 (3.47)

8. Secondary Outcome: Change in Quality of Life (QOL) and Caregiver Burden as Determined by the World Health Organization Quality of Life (WHOQOL-BREF) Questionnaire - Domain 2 (Psychological Health)
Description: Change in QOL/caregiver burden was assessed using the abbreviated WHOQOL-BREF. The WHOQOL-BREF measures 4 broad domains: Physical Health, Health, Social Relationships, and Environment. The questionnaire was completed by the parent/caregiver quantified the burden placed on the caregiver/family by the PWS disorder. For the Psychological Health domain (6 questions), responses were assigned to corresponding predefined scores ranging from 1-5 points. A mean overall Psychological Health score was calculated by summing the scores from 5 of the questions (#s 5, 6, 7, 11, and 19) and inverting the response value from Question #26 and adding it to the sum of the other 5 scores and dividing by the total number of questions (6). This result was multiplied by 4 to get a final Psychological Health domain score. Raw scoring ranges from 6-30; however, for purposes of this outcome measure change from baseline was reported. Positive values were associated with higher QOL and reduced caregiver burden.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | -0.500 (1.99) | -1.86 (3.90)

9. Secondary Outcome: Change in Quality of Life (QOL) and Caregiver Burden as Determined by the World Health Organization Quality of Life (WHOQOL-BREF) Questionnaire - Domain 3 (Social Relationships)
Description: Change in QOL and caregiver burden was assessed using the abbreviated WHOQOL-BREF. The WHOQOL-BREF measures 4 broad domains: Physical Health, Psychological Health, Social Relationships, and Environment. The questionnaire was completed by the parent/caregiver and quantified the burden placed on the caregiver/family by the PWS disorder. For the Social Relationships domain (3 questions), responses were assigned to corresponding predefined scores ranging from 1-5 points. A mean overall Social Relationships score was calculated by summing the 3 scores (#s 20, 21, and 22) and dividing by the total number of questions (3). This result was multiplied by 4 to get a final Social Relationships domain score. Social Relationships raw scoring ranges from 3-15; however, for purposes of this outcome measure change from baseline was reported. Positive values were associated with higher QOL and reduced caregiver burden.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | 0.00 (1.80) | 0.0714 (2.43)

10. Secondary Outcome: Change in Quality of Life (QOL) and Caregiver Burden as Determined by the World Health Organization Quality of Life (WHOQOL-BREF) Questionnaire - Domain 4 (Environment)
Description: Change in QOL and caregiver burden was assessed using the abbreviated WHOQOL-BREF. The WHOQOL-BREF is comprised of 26 items which measure 4 broad domains: Physical Health, Psychological Health, Social Relationships, and Environment. The questionnaire was completed by the parent/caregiver and quantified the burden placed on the caregiver/family by the PWS disorder. For the Environment domain (8 questions), responses were assigned to corresponding predefined scores ranging from 1-5 points. A mean overall Environment score was calculated by summing the scores from the 8 questions (#s 8, 9, 12, 13, 14, 23, 24, and 25) and dividing by the total number of questions (8). This result was multiplied by 4 to get a final Environmental domain score. Environment raw scoring ranges from 8-40; however, for purposes of this outcome measure change from baseline was reported. Positive values were associated with higher QOL and reduced caregiver burden.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 14 | 14
score on a scale | -0.0714 (1.86) | 0.571 (4.50)

11. Secondary Outcome: Change in Caregiver Strain
Description: Change in Caregiver Strain from baseline was assessed using the Caregiver Strain Questionnaire (CSQ). The CSQ is a 21-item measure of self-reported strain experienced by caregivers/families of youth with emotional problems. Responses to the CSQ are measured on a 5-point Likert scale measuring the impact of strain ranging from 1 = ("Not at all") to 5 = ("very much") for an overall possible scoring range of 21-105. For purposes of this outcome measure, a change in group mean score from baseline is summarized. A negative score is indicative of decreased caregiver/family strain from baseline; whereas, a positive score is indicative of increased caregiver/family strain from baseline.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: Data was unable to be collected from 2 participants in the matched Placebo study arm who withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | -1.32 (1.05) | -0.355 (1.35)

12. Secondary Outcome: Change in Aberrant Behavior
Description: Change in Aberrant Behavior from baseline was assessed using the Aberrant Behavior Checklist-Irritability 15-item subscale (ABC-I). The ABC-I subscale was completed by the caregiver on behalf of the child. At the suggestion of the FDA, the ABC-I subscale was included as a prospective assessment for suicidal ideation and behavior and inform investigators of trends toward increased irritability and disruptive behavior. ABC-I measures behavior on a 4-point severity scale where 0 = no problem at all, 1 = behavior is a problem but in a slight degree, 2 = problem is moderately serious, and 3 = problem is severe in degree, for an overall scoring range of 0-45. For purposes of this outcome, a change in group mean score from baseline is summarized. A negative ABC-I score is indicative of overall decreased irritability and disruptive behavior from baseline, whereas a positive ABC-I score is indicative of overall increased irritability and disruptive behavior from baseline.
Time Frame: From Randomization at Baseline until Endpoint at Week 8 (Change over 8 weeks)
Population: Data was unable to be collected from 2 participants in the matched Placebo study arm who withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | -5.33 (6.75) | -1.77 (5.95)

13. Secondary Outcome: Change in Salivary Oxytocin Concentration
Description: Change in Salivary Oxytocin concentration levels from baseline were to have been collected. Salivary samples were to have been collected using the Oragene-Discover collection kit (ORG-500). If able, participants were to have spit saliva directly into the collection tube during an in office or remote visit, and subsequently transported to the clinical site during visit and later processed and submitted for analysis. Change in group mean concentrations from baseline was to have been summarized by study arm using basic descriptive statistics. Increases in concentrations of salivary oxytocin are generally correlated with central nervous system effects and an improvement in these symptoms.
Time Frame: From Baseline until collections at 1 hour (Day 1), Week 4 and Week 8
Population: Due to challenges in collecting saliva samples from this population, participants were not able to provide enough saliva to allow for appropriate analysis. As such, samples were not obtained and data was unable to be collected.
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Clinical Global Impression Scale - Improvement (CGI-I)
Description: CGI-I is a clinician rated global measure of improvement that requires the clinician to assess how much the patient's illness has improved or worsened relative to baseline at the beginning of the intervention. The CGI-I consists of one query which is rated on a 7-point scale: "Compared to the patient's condition at admission [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment." Scores are summarized by study arm using basic descriptive statistics.
Time Frame: 8 weeks (measuring change over 8 weeks)
Population: Data was unable to be collected from 2 participants in the matched Placebo study arm who withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 2.93 (0.884) | 3.00 (1.000)

ADVERSE EVENTS:
Time Frame: Adverse event data for each subject was collected from baseline to completion of endpoint collection, 10 weeks total
Arm/Group | Experimental: Intranasal Oxytocin (IN-OXT) | Placebo Comparator: Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 7/15 | 13/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Intranasal Oxytocin (IN-OXT) (N=15) | Placebo Comparator: Matched Placebo (N=17)
Fatigue (General disorders) | 0 (0) | 3 (3)
Increased Irritability (Psychiatric disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aggressive Episode (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Strep Throat (Infections and infestations) | 0 (0) | 1 (1)
Nasal Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash - Upper Arms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Increased Episodes of Crying (Psychiatric disorders) | 1 (1) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Verbatim Term: Earache
Increased Speech Apraxia (Nervous system disorders) | 0 (0) | 1 (1)
Wet Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Sluggish (General disorders) | 0 (0) | 1 (1)
Hand, Foot, and Mouth Disease (Infections and infestations) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Exacerbated Skin Picking (Psychiatric disorders) | 0 (0) | 1 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Canker Sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Irritation Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Verbatim Term: Stomach Ache
Congestion (General) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03197662/Prot_SAP_000.pdf